CLINICAL TRIAL: NCT01491516
Title: A Pilot, Prospective, Non-Randomized Clinical Investigation of TELAMON P™ Implant With INFUSE® Bone Graft and the CD HORIZON® Spinal System for Posterior Lumbar Interbody Fusion in Patients With Symptomatic Degenerative Disc Disease
Brief Title: TELAMON P™ Implant/INFUSE® Bone Graft/CD HORIZON® Spinal System Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P01-07
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2011-12

CONDITIONS: Degenerative Disc Disease
Keywords: Lumbar degenerative disc disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Investigational (Experimental)
  Interventions: Device: TELAMON P™ /INFUSE® Bone Graft/CD HORIZON® Spinal System

INTERVENTIONS:
Device: TELAMON P™ /INFUSE® Bone Graft/CD HORIZON® Spinal System — The TELAMON P™/INFUSE™ Bone Graft Implant in conjunction with the CD HORIZON® Spinal System for single level lumbar fusion from L1 to S1
  Other Names: PEEK OPTIMA™ LT

SUMMARY:
The purpose of this pilot study is to evaluate the feasibility of the implant ( TELAMON P™ Implant/INFUSE Bone Graft System used in conjunction with the CD HORIZON® Spinal System) as a method of facilitating lumbar spinal fusion utilizing a posterior surgical approach in patients with symptomatic degenerative disc disease. The safety and effectiveness of the implant will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Has degenerative disc disease as noted by back pain of discogenic origin, with or without leg pain, with degeneration of the disc confirmed by patient history and radiographic studies to include one or more of the following:

   * instability (defined as angulation >= 5° and/or translation >= 4mm, based on flexion/extension radiographs);
   * osteophyte formation;
   * decreased disc height;
   * thickening of ligamentous tissue;
   * disc degeneration or herniation; and/or
   * facet joint degeneration.
2. Has preoperative Oswestry score >= 30.
3. Has preoperative back pain score of >= 25 based on the Preoperative Back and Leg Pain Questionnaire (intensity and duration).
4. Has no greater than Grade 1 spondylolisthesis utilizing Meyerding's Classification (Meyerding, HW, 1932).
5. Requires fusion of a single level disc space from L 1 to S 1.
6. Is at least 18 years of age, inclusive, at the time of surgery.
7. Has not responded to non-operative treatment for a period of 6 months.
8. If of child-bearing potential, patient is non-pregnant, non-nursing, and agrees to not get pregnant for 1 year following surgery.
9. Is willing and able to comply with the study plan and sign the Patient Informed Consent Form.

Exclusion Criteria:

1. Has primary diagnosis of a spinal disorder other than degenerative disc disease with Grade 1 or less spondylolisthesis at the involved level.
2. Had previous spinal fusion surgical procedure at the involved level.
3. Requires spinal fusion at more than one lumbar level.
4. Has a condition which requires postoperative medications that interfere with fusion, such as steroids or prolonged use of nonsteroidal anti-inflammatory drugs excluding routine peri-operative nonsteroidal anti-inflammatory drugs. This does not include low dose aspirin for prophylactic anticoagulation.
5. Has been previously diagnosed with osteopenia or osteomalacia.
6. Has any of the following that may be associated with a diagnosis of osteoporosis (if "Yes" to any of the below risk factors, a dual x-ray absorptiometry (DEXA) Scan will be required to determine eligibility).

   1. Postmenopausal Non-Black female over 60 years of age and weighs less than 140 pounds.
   2. Postmenopausal female that has sustained a non-traumatic hip, spine, or wrist fracture.
   3. Male over the age of 70.
   4. Male over the age of 60 that has sustained a non-traumatic hip or spine fracture. If the level of BMD is a T score of -3.5 or a T score of -2.5 with vertebral crush fracture, the patient is excluded from the study.
7. Has presence of active malignancy or prior history of malignancy, except for basal cell carcinoma of the skin.
8. Has an overt or active bacterial infection, either local or systemic.
9. Has a documented titanium, titanium alloy, tantalum, tantalum alloy, or polyetheretherketone allergy or intolerance.
10. Is mentally incompetent. If questionable, obtain psychiatric consult.
11. Has a Waddell Signs of Inorganic Behavior score of 3 or greater.
12. Is a prisoner.
13. Is an alcohol and/or drug abuser as defined by currently undergoing treatment for alcohol and/or drug abuse.
14. Has received drugs which may interfere with bone metabolism within two weeks prior to the planned date of spinal fusion surgery (e.g., steroids or methotrexate), excluding routine perioperative antiinflammatory drugs.
15. Has a history of any autoimmune disease (e.g. Systemic Lupus Erythematosus or Dermatomyositis) .
16. Has a history of exposure to injectable collagen or silicone implants.
17. Has a history of hypersensitivity to protein pharmaceuticals (e.g. monoclonal antibodies or gamma globulins) or collagen.
18. Has received treatment with an investigational therapy (device and/or pharmaceutical) within 28 days prior to implantation surgery or such treatment is planned during the 16 weeks following the investigational treatment.
19. Has received any previous exposure to any/all BMP's of either human or animal extraction.
20. Has a history of allergy to bovine products or a history of anaphylaxis.
21. Has history of any endocrine or metabolic disorder known to affect osteogenesis (e.g., Paget's disease, renal osteodystrophy, Ehlers-Danlos syndrome, or osteogenesis imperfecta).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-07; Primary Completion 2008-04 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Overall Success | 24 month
  A patient will be considered an overall success if all of the following conditions are met:
  1. fusion;
  2. pain/disability (Oswestry) success;
  3. neurological status success;
  4. no serious adverse event classified as "implant associated" or "implant/surgical procedure associated";
  5. no additional surgical procedure classified as a "failure".

SECONDARY OUTCOMES:
Disc Height Measurement | 24 month
General Health Status (SF-36) | 24 month
Pain Status (back pain, leg pain) | 24 month
Patient Satisfaction | 24 month
Patient Global Perceived Effect | 24 month